CLINICAL TRIAL: NCT04432701
Title: Which is the Better Choice for Extubation in Pediatric Patients: Proactive or Passive?
Brief Title: Extubation in Pediatric Patients: Proactive or Passive?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A/P extubation
Record Dates: First submitted 2020-05-03; First posted 2020-06-16 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Cough; Tracheal Extubation
Keywords: passive; proactive; extubation; respiratory complication
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Active Comparator): children were extubated in a light plane of anesthesia, when they are still asleep or have swallowing reflex.
  Interventions: Behavioral: proactive extubation
- group B (No Intervention): Tracheal extubation was performed when the patient regained consciousness, facial grimace, spontaneous eye opening, and purposeful arm movement.

INTERVENTIONS:
Behavioral: proactive extubation — when children is breathing spontaneously and adequately in PACU,endotracheal tube was removed directly
  Arms: group A

SUMMARY:
Smooth extubation process can reduce the complications in recovery time. This study aimed to investigate what is the better time to extubation when children is breathing spontaneously and adequately: waiting until children have movements or wakefulness (passive extubation）or removing endotracheal tube directly (proactive tracheal extubation).

DETAILED DESCRIPTION:
This is a randomized, controlled cross-over trial. The hypothesis of this study is that the different extubation protocol can impact recovery quality in children in post-anaesthesia care unit (PACU). Patients aged 3-7 years were randomized into two equal groups: proactive extubation (Group A) and passive extubation. At the end of surgery, sevoflurane was turned off and patients all delivered into PACU for recovery. Patient was positioned on his or her lateral side. The ventilation was switched to positive airway pressure (CPAP) mode once the patients regained spontaneous respiration. After spontaneous breathing turn to regular and sufficient（tidal volume >6-8 ml/kg, respiratory rate >10 times per minutes , end tidal carbon dioxide concentration >7.19 mmHg）, the trachea tube could be removed. In Group A, patients were extubated in a light plane of anesthesia, when they are still asleep or have swallowing reflex. In Group B, tracheal extubation was performed when the patient regained consciousness, facial grimace, spontaneous eye opening, and purposeful arm movement. After extubation, 2 L/min oxygen was administered with Venturi face mask for 10 min in both groups. Patients were transported to the ward until they breathed air with a patent airway. The extubation time, recovery characteristics and respiratory complication were recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status aged 3-7 years

Exclusion Criteria:

* a suspected difficult airway reactive airway disease, recent upper respiratory tract infection gastrointestinal reflux obesity (body mass index>30 kg/m2

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Coughing | at the time of extubation within 1 minute
  1 if a single cough occurred and saturation by pulse oximetry (SpO2) ≥95%; 2 if multiple coughs occurred and SpO2 ≥95%; 3 if multiple coughs occurred and SpO2 <95%; and 4 if multiple coughs occurred, SpO2 <95%, and coughing required administration of i.v . medication.
Respiratory complications | During the time when patients stayed in PACU after extubation, an average of 45 min
  the number of patients who had gagging, clenched teeth, gross purposeful movements, breath holding, laryngospasm, or desaturation to SpO2<90%
Time to spontaneous eye opening | The time from PACU arrival to spontaneous eye opening, an average of 45 min
  Time to spontaneous eye opening
Time to discharge from PACU | The time from patients arrived PACU to who was decided to discharge from PACU，an average of 1 hour
  Time to discharge from PACU

SECONDARY OUTCOMES:
Time to extubation | The time from PACU arrival to tracheal extubation, an average of 30 min
  The time of extubation after surgery
End-tidal concentration of minimum effective alveolar anesthetic concentration | The time before patients were decided to extubate, within 1 minute
  In percentage
Age | 6 hours before intervention
  In years
Weight | 6 hours before intervention
  In kilograms
Height | 6 hours before intervention
  In meters
Systolic blood pressure | 5 minutes before extubation
  Hemodynamic parameter
Systolic blood pressure | 1 minute after extubation
  Hemodynamic parameter
Systolic blood pressure | 5 minutes after extubation
  Hemodynamic parameter
Diastolic blood pressure | 5 minutes before extubation
  Hemodynamic parameter
Diastolic blood pressure | 1 minute after extubation
  Hemodynamic parameter
Diastolic blood pressure | 5 minutes after extubation
  Hemodynamic parameter
Heart rate | 5 minutes before extubation
  hemodynamic parameter
Heart rate | 1 minute after extubation
  hemodynamic parameter
Heart rate | 5 minutes after extubation
  hemodynamic parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsukamoto M, Hitosugi T, Yokoyama T. Comparison of recovery in pediatric patients: a retrospective study. Clin Oral Investig. 2019 Sep;23(9):3653-3656. doi: 10.1007/s00784-019-02993-y. Epub 2019 Jul 4. PMID 31273527
- [Background] Bidwai AV, Bidwai VA, Rogers CR, Stanley TH. Blood-pressure and pulse-rate responses to endotracheal extubation with and without prior injection of lidocaine. Anesthesiology. 1979 Aug;51(2):171-3. doi: 10.1097/00000542-197908000-00020. No abstract available. PMID 453622
- [Background] Valley RD, Freid EB, Bailey AG, Kopp VJ, Georges LS, Fletcher J, Keifer A. Tracheal extubation of deeply anesthetized pediatric patients: a comparison of desflurane and sevoflurane. Anesth Analg. 2003 May;96(5):1320-1324. doi: 10.1213/01.ANE.0000058844.77403.16. PMID 12707126
- [Result] Gonzalez RM, Bjerke RJ, Drobycki T, Stapelfeldt WH, Green JM, Janowitz MJ, Clark M. Prevention of endotracheal tube-induced coughing during emergence from general anesthesia. Anesth Analg. 1994 Oct;79(4):792-5. doi: 10.1213/00000539-199410000-00030. No abstract available. PMID 7943794
- [Result] Fan Q, Hu C, Ye M, Shen X. Dexmedetomidine for tracheal extubation in deeply anesthetized adult patients after otologic surgery: a comparison with remifentanil. BMC Anesthesiol. 2015 Jul 23;15:106. doi: 10.1186/s12871-015-0088-7. PMID 26202786
- [Result] Inomata S, Yaguchi Y, Taguchi M, Toyooka H. End-tidal sevoflurane concentration for tracheal extubation (MACEX) in adults: comparison with isoflurane. Br J Anaesth. 1999 Jun;82(6):852-6. doi: 10.1093/bja/82.6.852. PMID 10562778